CLINICAL TRIAL: NCT06671457
Title: Model-Driven Individualized Transcranial Direct Current Stimulation for the Treatment of Insomnia Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhen Wang (Other)
Responsible Party: Sponsor-Investigator, Zhen Wang, vice president, Shanghai Mental Health Center
Organization: Shanghai Mental Health Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMHC-ISM-002
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Insomnia
Keywords: insomnia; transcranial direct current stimulation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Group (Experimental): To optimize stimulation parameters, electromagnetic modeling and parameter space scanning of the participant's brain are conducted. The specific method includes performing MRI scans before stimulation. MRI structural data is then used to create individualized models of the participant's brain and simulate the electromagnetic fields within biological tissues. High-density EEG is collected during the participant's sleep state, using a 256-channel stimulation-recording device (MagStim EGI, GTEN 200) to record EEG changes induced by stimulation across multiple brain regions. The type of electrical stimulation is cathodal direct current stimulation, targeting brain regions with an intensity equivalent to the traditional 2mA single-channel current, with each electrode not exceeding 200μA. Target brain regions for stimulation include the dorsolateral prefrontal cortex (DLPFC), orbitofrontal cortex (OPFC), medial prefrontal cortex (mPFC), and posterior cingulate cortex (PCC). Changes in brain
  Interventions: Device: Active transcranial direct current stimulation
- Sham Group (Sham Comparator): In the sham stimulation group, the placement of the tDCS electrodes is identical to that of the active stimulation group. After the stimulation begins, the current gradually increases over 15 seconds. However, upon reaching the therapeutic current level, it immediately begins to decrease, lowering to 0 mA within 15 seconds and remaining at 0 mA throughout the rest of the session. During the last 15 seconds of the stimulation, there is another gradual decrease in current to 0 mA. This approach creates a similar subjective sensation to the real stimulation, making it difficult for participants to discern which type of electrical stimulation they are receiving.
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Active transcranial direct current stimulation — The intervention uses transcranial direct current stimulation (tDCS). The targeted brain regions are identified by conducting simultaneous fMRI-EEG data collection and sleep staging, comparing fMRI data between wakefulness and sleep states. Brain regions that show differences are calculated as potential targets for electrical stimulation. If no differentiated regions are found in a participant, specific areas are chosen based on individualized modeling results from previous experiments, targeting areas such as the dorsolateral prefrontal cortex (DLPFC), orbitofrontal cortex (OPFC), medial prefrontal cortex (mPFC), and posterior cingulate cortex (PCC). Two regions are selected within each brain area for parameter scanning (with each stimulation lasting 10 seconds and EEG data recorded 10 seconds before and after stimulation).
  In our prior studies, we observed a decrease in EEG microstate complexity during sleep, with electrical stimulation influencing this complexity reduction to some
  Arms: Active Group
Device: Sham transcranial direct current stimulation — In the sham stimulation group, the placement of the tDCS electrodes is identical to that of the active stimulation group. After the stimulation begins, the current gradually increases over 15 seconds. However, upon reaching the therapeutic current level, it immediately begins to decrease, lowering to 0 mA within 15 seconds and remaining at 0 mA throughout the rest of the session. During the last 15 seconds of the stimulation, there is another gradual decrease in current to 0 mA. This approach creates a similar subjective sensation to the real stimulation, making it difficult for participants to discern which type of electrical stimulation they are receiving.
  Arms: Sham Group

SUMMARY:
This study is designed to evaluate the efficacy and to explore the best individualized stimulus paradigm of transcranial Electrical Stimulation for insomnia patients.

DETAILED DESCRIPTION:
This study employs a randomized double-blind placebo-controlled design, with blinding applied to both the assessors and patients, while the therapists remain unblinded. A total of 40 patients with insomnia disorders meeting the inclusion criteria were recruited from the Shanghai Mental Health Center and randomly assigned to either the tDCS active stimulation group or the tDCS sham stimulation group, with 20 patients in each group. All patients underwent clinical assessments, magnetic resonance imaging (MRI) scans, and high-density electroencephalogram (EEG) parameter collections at baseline. Based on the MRI structural images and high-density EEG parameters, individualized modeling was conducted to determine specific stimulation parameter schemes (stimulation sites, stimulation intensity, and electrode placement methods). Detailed modeling methods and selection of stimulation parameters can be found in the intervention methods section. Stimulation was carried out for a total of 2 weeks, with one session per day on weekdays, totaling 10 sessions, each lasting thirty minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years;
2. Meets the diagnostic criteria for insomnia disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
3. Has not taken psychiatric medications in the 8 weeks prior to enrollment or has been on stable psychiatric medication for 8 weeks (excluding benzodiazepines);
4. Insomnia severity as indicated by an ISI score > 10;
5. Minimum education level of junior high school or above.

Exclusion Criteria:

1. Past or current diagnosis of disorders other than insomnia disorder, anxiety disorder, or depressive disorder according to DSM-5;
2. Currently using benzodiazepines as sleep aids;
3. Moderate to severe anxiety or depression (HAMD-17 score > 16 or HAMA score > 24);
4. Patients with obstructive sleep apnea syndrome;
5. Previous treatment with ECT, rTMS, tES, or cognitive behavioral therapy for insomnia disorder;
6. Severe physical illnesses or any condition that may induce seizures or intracranial hypertension, including cardiovascular or respiratory diseases;
7. History of neurological disorders (e.g., epilepsy, cerebrovascular accidents) or history of brain injury or brain surgery;
8. Presence of implantable medical devices such as intracranial stents, cardiac pacemakers, coronary stents, or cochlear implants;
9. Severe negative thoughts or high suicide risk;
10. Pregnant or planning to conceive in the near future.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index change | The study endpoint is set at 2 weeks after the end of treatment
  The change of the Insomnia Severity Index (ISI) score.The scale consists of 7 items, scored on a 5-point Likert scale ranging from 0 to 4 for each item, with a total score ranging from 0 to 28. Higher scores indicate more severe insomnia.

SECONDARY OUTCOMES:
Insomnia Severity Index score change | after tDCS intervention and 4 weeks post-intervention
  the change in the Insomnia Severity Index (ISI) score after tDCS intervention and 4 weeks post-intervention.
response/remission rate | After tDCS intervention, 2 weeks post-intervention, and 4 weeks post-intervention
  Treatment effectiveness is defined as a reduction of more than 7 points in the Insomnia Severity Index (ISI) score post-treatment. Clinical remission is defined as a total ISI score of less than 8 points.
Sleep onset latency, sleep efficiency, and nighttime sleep duration (as defined by the sleep diary). | After tDCS intervention and 2 weeks post-tDCS intervention
  Changes in sleep onset latency, sleep efficiency, and nighttime sleep duration after tDCS intervention and 2 weeks post-tDCS intervention.
Hamilton Depression Rating Scale-17 change | After tDCS intervention, 2 weeks post-tDCS intervention, and 4 weeks post-intervention
  Hamilton Depression Rating Scale 17 score change after tDCS intervention, 2 weeks post-tDCS intervention, and 4 weeks post-intervention. For the HDRS17 , a score of 0-7 is generally accepted to be within the normal Hamilton Depression Rating Scale (HDRS) range (or in clinical remission), while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial. Higher scores indicate more severe depression.
Hamilton Anxiety Rating Scale Change | After tDCS intervention, 2 weeks post-tDCS intervention, and 4 weeks post-intervention
  Hamilton Anxiety Rating Scale score change after tDCS intervention, 2 weeks post-tDCS intervention, and 4 weeks post-intervention.Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD,MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided